CLINICAL TRIAL: NCT02221427
Title: The Labour Progression Study, a Cluster Randomised Trial on Labour Progression for First Time Mothers
Acronym: LAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Stine Bernitz, Midwife, PhD, Ostfold Hospital Trust
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: LAPS3293
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Caesarean Sections; Augmentation With Oxytocin; Labour Dystocia
Keywords: First time mothers; Labour progression; Prolonged labour; Oxytocin; Mode of delivery; Maternal birth outcome; Neonatal birth outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Static labour progression curve (F) (Active Comparator): Guideline with the following expected labour progression: if the cervix dilates at least 1 centimetre per hour assessed after 4 hours. Labour dystocia is diagnosed if progression proceeds slower than this definition throughout the active phase of the first stage of labour. Labour dystocia in the second stage of labour is diagnosed if lasting longer than two hours, three hours for women with epidurals or if the expulsion phase lasts longer than 60 minutes.
  Interventions: Other: Static labour progression curve (F)
- Dynamic progression curve (Z) (Experimental): Guideline which takes into account the dilatation of the cervix on admission and calculates the expected progression during the active phase of the first stage of labour based on this finding. Labour dystocia in the second stage of labour is diagnosed if lasting longer than two hours and 45 minutes, three hours and 30 minutes for women with epidurals or if the expulsion phase lasts longer than 60 minutes.
  Interventions: Other: Dynamic progression curve

INTERVENTIONS:
Other: Dynamic progression curve — Guideline which takes into account the dilatation of the cervix on admission and calculates the expected progression during the active phase of the first stage of labour based on this finding. Labour dystocia in the second stage of labour is diagnosed if lasting longer than two hours and 45 minutes, three hours and 30 minutes for women with epidurals or if the expulsion phase lasts longer than 60 minutes. This guideline is based on the labour progression curve by Zhang.
  Other Names: Zhang's progression curve
  Arms: Dynamic progression curve (Z)
Other: Static labour progression curve (F)
  Arms: Static labour progression curve (F)

SUMMARY:
The purpose of this study is to evaluate if the rate of emergency caesarean section can be reduced if adhering to a dynamic labour progression curve compared to a static progression curve for first time mothers without jeopardising maternal and neonatal outcomes

DETAILED DESCRIPTION:
1. Introduction The increasing rate of emergency caesarean sections in developed countries is of great concern as it is associated with adverse outcomes for mother and infant. The rate of caesarean sections for first time mothers with a singleton foetus in a vertex position and spontaneous onset of labour at term has increased from 5.7 % to 9.2 % in Norway. The most common indication for emergency caesarean sections is Labour dystocia, even if there is no consensus on criteria for the diagnosis.

   Labour dystocia is characterised by abnormally slow progress of labour and is among the most common challenges of birth care especially in first time mothers. When the labour progression is assessed to be prolonged according to current guidelines, labour dystocia is treated by amniotomy followed by oxytocin infusion to augment uterus contractions. Oxytocin is a potent drug and classified by the Institute for Safe Medication Practices in the USA as one of 12 medications which is "bearing heightened risk of harm".

   In Norway the guidelines for expected progression of labour is based on modifications of Friedman's curve of cervical dilatation, a linear labour progression curve developed in 1953. Contemporary research by Zhang shows that the dilatation of the cervix can be substantially slower than earlier expected, especially at an early stage of labour.

   Hypothesis: By adhering to the guideline for labour progression presented by Zhang, the rate of emergency caesarean sections in first time mothers will decrease compared to adhering to the guideline for labour progression based on a modified Friedman's curve, without jeopardising the maternal and neonatal outcomes.
2. Background and status of knowledge Traditionally the labour process is divided in two stages; the first stage and the second stage. The first stage is divided in two phases; the latent phase and the active phase, the latent phase is defined from onset of labour until the cervix is dilated four centimetres with 3-4 painful contractions per ten minutes. The active phase is defined from a cervix dilatation of four centimetres until fully dilated. The second stage is divided in two phases; the deceleration phase where the baby's head is decelerating towards the pelvic floor and the expulsion phase where the mother is actively pushing the baby out.

   To visualize the progression of labour, the status of the cervix dilatation is traditionally measured and recorded throughout labour on a graphic curve often called a partogram. The partogram is widely used internationally and facilitates that midwives' and doctors' can monitor labour progression, and together with criteria for labour dystocia, consequently carry out necessary interventions.

   In 1954 Dr. Friedman presented the first progression curve based on examination of 100 first time mothers. Friedman's curve has been widely adopted and applied in practice internationally for almost 60 years. In 2002 Dr. Zhang presented a new labour curve based on labour data from 1329 low-risk women. Zhang's findings were confirmed in a large cohort of 26,838 women in 2010.

   Zhang's labour curve differs markedly from the Friedman's curve in that the cervix dilates substantially slower, especially before reaching six centimetres of dilatation, nor is the distinct deflection of the curve between nine and ten centimetres in Friedman's curve found in Zhang's curve. These findings may suggest that the diagnostic criteria for labour dystocia are too stringent following Friedman's curve in contemporary birth care.

   A new guideline for normal birth progression is developed according to Zhang's curve and contemporary research findings. The new guideline differs from the existing ones by not expecting a linear progression and by defining the progression to be normal if the speed of cervical dilatation is within the 95 percentile of the duration in Zhang's material. Active labour is defined when the cervical dilatation is 4 centimetres or more until the baby is born. In this dynamic labour curve, labour dystocia is defined if time from 4 to 5 cm exceeds six hours and 30 minutes, if time from 5 to 6 cm exceeds three hours and 15 minutes, if time from 6 to 7 cm exceeds two hour and 15 minutes, if time from 7 to 8 cm exceeds one hour and 30 minutes, if time from 8 to 9 cm exceeds one hour and 30 minutes or if time from 9 to 10 cm exceeds one hour and 45 minutes.

   New knowledge and competence on labour progression may result in a new guideline allowing low-risk labours to proceed without unnecessary interventions which will benefit the population both medically and economically.
3. Design and implementation To evaluate if our hypothesis is true, a cluster randomised trial will be conducted. The objective is to include birth care units by randomising them to adhere to either of the two guidelines in active labour; F (Standard care according to Friedman's guideline) or Z; (Experimental care according to Zhang's guideline) F = Guideline with the following expected labour progression: if the cervix dilates at least 1 centimetre per hour assessed after 4 hours. Labour dystocia is diagnosed if progression proceeds slower than this definition throughout the active phase of the first stage of labour. Labour dystocia in the second stage of labour is diagnosed if lasting longer than two hours, three hours for women with epidurals or if the expulsion phase lasts longer than 60 minutes. This guideline is based on an interpretation of Friedman's expected progression of labour.

Z = Guideline which takes into account the dilatation of the cervix on admission and calculates the expected progression during the active phase of the first stage of labour based on this finding. Labour dystocia in the second stage of labour is diagnosed if lasting longer than two hours and 45 minutes, three hours and 30 minutes for women with epidurals or if the expulsion phase lasts longer than 60 minutes. This guideline is based on the labour progression curve by Zhang.

Fourteen clusters will be included. The choice of cluster randomising, is due to the risk of contamination if randomised on an individual level. Key elements to specify regarding allocation of treatment are: The method of generating the allocation sequence is computer-generated, the allocation ratio is equal to one, and the type of randomisation is restricted and the factors "size of birth care unit" and "prior rates of caesarean sections for first time mothers with a singleton foetus in a vertex position, in spontaneous onset of labour at term" will be used for stratification.

The randomisation process will be performed through a central computer assisted programme. The trial will be conducted according to the CONSORT statement for planning and implementation of cluster randomised trials.

All clusters will receive a concise edition of the trial protocol and sign the cooperation agreement.

Each cluster must also provide one dedicated person (local coordinator) responsible for the trial during the inclusion period. The local coordinator is responsible for recruitment and inclusion of participants, monitoring the entries in a web-Case Report Form (web-CRF), record control of each participant and is responsible for the implementation of the trial.

For each included cluster, all the following criteria must be met: Birth care units that are willing to adhere to the guidelines in the trial period and who consider that they have the capacity to participate both logistical and practical. The size of the birth care units should be more than 500 deliveries per year to secure a reasonable inclusion period.

Statistical methods and data analysis: The determination of the sample size is based on a power calculation with the least occurring outcome; emergency caesarean section, which is 9.2 % in the study population (p1). Further, we expect that the emergency caesarean section rate will be 6.7 % (p2) which id a 25 % reduction, when using the new guideline. With a chosen significance level of 0.05, a power of 80 % and p1=9.2 % and p2=6.9 %, we will have to include at least 14 clusters and 6582 individuals. As we are testing a new guideline, blinding of care givers is not possible. The statistician will perform analyses blinded to the participant's affiliation to the groups as a control of the analysis.

Analysis: The difference between the randomized groups will be presented with a Risk Ratio (RR) and a 95 % confidence interval (95% CI). For dichotomous efficacy variables a significance test taking into account the cluster structure of the data, will be used. For continuous data an independent sample t-test will be used. Statistical analysis will be conducted using STATA version 10.1 StataCorp, Texas, //845 USA and SPSS version 18. The analyses will be conducted according to the principle of intention to treat.

Implementation All first time mothers with a singleton foetus in a vertex position, in spontaneous onset of labour at term will adhere to the labour progression guideline that the cluster is randomised to.

All eligible participants will receive written information about the trial when called for routine ultrasound control, at the routine ultrasound control or at the labour ward. They will be asked to sign an informed consent permitting her data to be included in the analyses, and to answer an on-line questionnaire about her childbirth experience.

Safety assessment: All women in both arms will be cared for and monitored according to the procedures at each birth care unit. Necessary interventions due to the mother's or the fetus' needs, will be conducted regardless of the allocated guideline for labour progression.

Web-Case Report Form: Due to different systems for electronic medical records and due to additional handwritten records, a web based Case Report Form (web-CRF) is being designed by the Unit of Applied Clinical Research at the Faculty of Medicine at the Norwegian University of Science and Technology, NTNU. The web-CRF is transferable to the analytical tools; STATA and SPSS. The local coordinators will ensure that the data required by the protocol is entered de-identified into the web-CRF. The local coordinators are also responsible for assuring that data entered into the web-CRF is complete, accurate, and that entry is performed in a timely manner. The signature of the local coordinators will attest to the accuracy of the data on each web-CRF.

Consecutively assessments will be recorded in the electronic journal throughout labour, assessments recorded on the printed version of the partogram will be transmitted to the web-CRF at each birth care unit. Assessments to be recorded throughout labour are e.g.: Cervix status on admission (in centimetres), results of regularly vaginal exploration, the use of oxytocin, pain relief and additional interventions.

The trial manager shall arrange for the secure retention of the participant identification and the code list. Participant files shall be kept for the maximum period of time permitted by each birth care unit. The trial documentation (web-CRF, Site File etc.) shall be retained and stored during the trial and for 10 years after trial closure. All information concerning the trial will be stored in a safe place inaccessible to unauthorized personnel.

Investigator Delegation Procedure: The trial manager is responsible for making and updating a "delegation of tasks" listing all the involved co-workers and their role in the project. The principle investigators will ensure that appropriate training relevant to the study is given to the staff, and that any new information of relevance to the performance of this trial is forwarded to the staff involved.

All significant protocol deviations will be recorded and reported in the Clinical Study Report (CSR).

If it is necessary for the study protocol to be amended, the amendment and/or a new version of the trial protocol (Amended Protocol) must be notified to and approved by the Competent Authority and the Ethics Committees according to EU and national regulations.

Audit and Inspections: Authorized representatives of a Competent Authority and Ethics Committee may visit the centres to perform inspections, including source data verification. The purpose of an inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded, analysed, and accurately reported according to the protocol, Good Clinical Practice, and any applicable regulatory requirements. The principal investigators will ensure that the inspectors and auditors will be provided with access to source data/documents.

Publication policy: All personnel who have contributed significantly with the planning and performance of the study according to the Vancouver convention 1988 may be included in the list

Ethical and regulatory requirements: The trial will be conducted in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with Good Clinical Practice and applicable regulatory requirements. Registration of participant's data will be carried out in accordance with national personal data laws. The protocol, including the patient information and informed consent form to be used, is approved by the ethics committee in Norway: 2013/1862/REK sør-øst. The principal investigator is responsible for informing the ethics committee of any serious and unexpected adverse events and/or major amendments to the protocol as per national requirements.

The protocol must be approved by the management at the birth care units before commencement of the trial. The protocol will also be registered in www.clinicaltrials.gov before enrollment of participants.

ELIGIBILITY:
Inclusion Criteria:

* Robson group I:First time mothers with a singleton foetus in a vertex position, in spontaneous onset of labour between gestational week 37-42

Exclusion Criteria:

* Robson groups 2-10

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6582 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of emergency caesarean section | 14 months

SECONDARY OUTCOMES:
The use of oxytocin for augmenting uterus contractions | 14 months
  The rate of women augmented with oxytocin including indication for initiating oxytocin infusion, cervical dilatation at onset of augmentation and length of augmentation

OTHER OUTCOMES:
The rate of instrumental vaginal deliveries | 14 months
  The rate of both vacuum extractions and forceps deliveries
The rate of artificial rupture of membranes (amniotomy) | 14 months
The rate of electronic fetal monitoring | 14 months
  Electronic fetal monitoring including cardio tocography (CTG) both with and without ST analysis (STAN) will be recorded
The rate of epidural analgesia | 14 months
The rate of episiotomies | 14 months
The rate of anal sphincter injuries | 14 months
The rate of labour dystocia | 14 months
  The rate of prolonged labour according to allocated guideline for labour progression
Postpartum haemorrhage | 14 months
  The rate of postpartum haemorrhage of more than 1000 ml and the rate of blood transfusions post partum
Apgar scores | 14 months
  The rate of apgar scores less or equal to 7 after 10 minutes post partum
Ph in the umbilical artery | 14 months
The rate of transfers of neonates to the Neonatal Intensive Care Unit | 14 months
  The rate of transfers of neonates within two hours post partum
The mean duration of labour | 14 months
  The duration of labour in all phases of labour and in total
• Mean score of women's experience with child birth (measured by :"The Childbirth Experience Questionnaire, CEQ" | 14 months
  Four weeks after birth all Robson group I women will receive a request to complete an online questionnaire regarding birth experience, the Childbirth Experience Questionnaire CEQ

CONTACTS AND LOCATIONS:
Overall Officials: Stine Bernitz, PhD, Principal Investigator — Ostfold Hospital Trust
Locations (1):
- Østfold Hospital Trust, Fredrikstad, Østfold fylke, Norway

REFERENCES:
- [Derived] Husby AE, Simpson MR, Dalbye R, Larsen M, Vanky E, Lovvik TS. Childbirth experiences in women with polycystic ovary syndrome: A cohort study. Acta Obstet Gynecol Scand. 2024 Jun;103(6):1092-1100. doi: 10.1111/aogs.14800. Epub 2024 Feb 17. PMID 38366810
- [Derived] Bernitz S, Dalbye R, Zhang J, Eggebo TM, Froslie KF, Olsen IC, Blix E, Oian P. The frequency of intrapartum caesarean section use with the WHO partograph versus Zhang's guideline in the Labour Progression Study (LaPS): a multicentre, cluster-randomised controlled trial. Lancet. 2019 Jan 26;393(10169):340-348. doi: 10.1016/S0140-6736(18)31991-3. Epub 2018 Dec 20. PMID 30581039
- [Derived] Bernitz S, Dalbye R, Oian P, Zhang J, Eggebo TM, Blix E. Study protocol: the Labor Progression Study, LAPS - does the use of a dynamic progression guideline in labor reduce the rate of intrapartum cesarean sections in nulliparous women? A multicenter, cluster randomized trial in Norway. BMC Pregnancy Childbirth. 2017 Nov 13;17(1):370. doi: 10.1186/s12884-017-1553-8. PMID 29132336